CLINICAL TRIAL: NCT07365033
Title: Effectiveness of Eccentric Training With Blood Flow Restriction Therapy Versus Resistance Training in Patients With Lateral Epicondylitis
Brief Title: Eccentric Exercise With Blood Flow Restriction vs Resistance Training for Lateral Epicondylitis
Acronym: BFR-ET LE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nimra Rafiq (Other)
Responsible Party: Sponsor-Investigator, Nimra Rafiq, principal investigator, University of Lahore
Organization: University of Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB/25/15/03/28
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Lateral Epicondylitis
Keywords: Lateral Epicondylitis; Blood Flow Restriction Therapy; Eccentric Training; Resistance Training,
MeSH Terms: conditions — Tennis Elbow | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group A (Experimental): The interventional group will receive eccentric wrist extensor exercises combined with blood flow restriction therapy, using a pneumatic cuff inflated to 50-60% limb occlusion pressure. Exercises will be performed at 20-30% 1-RM using a 30-15-15-15 repetition protocol, emphasizing slow controlled eccentric contractions. Sessions will be conducted three times weekly for 8 weeks, totaling 24 supervised sessions.
  Interventions: Behavioral: interventional group A
- Control group B (Active Comparator): The control group will undergo a heavy slow resistance training protocol, involving wrist extensor exercises performed at 70-85% of 1-RM, with slow concentric and eccentric phases (3 seconds each). Participants will complete 3-4 sets of 6-8 repetitions, with adequate rest intervals, following the same session frequency and duration as the intervention group.
  Interventions: Behavioral: control group b

INTERVENTIONS:
Behavioral: interventional group A — The interventional group will receive eccentric wrist extensor exercises combined with blood flow restriction therapy, using a pneumatic cuff inflated to 50-60% limb occlusion pressure. Exercises will be performed at 20-30% 1-RM using a 30-15-15-15 repetition protocol, emphasizing slow controlled eccentric contractions. Sessions will be conducted three times weekly for 8 weeks, totaling 24 supervised sessions.
  Other Names: blood flow resistance training
  Arms: interventional group A
Behavioral: control group b — The control group will undergo a heavy slow resistance training protocol, involving wrist extensor exercises performed at 70-85% of 1-RM, with slow concentric and eccentric phases (3 seconds each). Participants will complete 3-4 sets of 6-8 repetitions, with adequate rest intervals, following the same session frequency and duration as the intervention group.
  Other Names: resistance training
  Arms: Control group B

SUMMARY:
This randomized controlled trial aims to compare the effectiveness of eccentric training combined with blood flow restriction (ECC+BFR) versus heavy slow resistance (HSR) training in patients with chronic lateral epicondylitis. The study will recruit 40 participants (accounting for 10% attrition), aged 25-45 years, from Sakina Memorial Hospital Sheikhupura and University of Lahore Teaching Hospital using convenience sampling. Participants will be randomly allocated into two groups: an interventional group receiving ECC+BFR and a control group undergoing HSR training. Both interventions will be administered three times per week for 8 weeks under professional supervision. Outcome measures including pain intensity (NPRS), patient-specific functional performance (PSFS), muscle strength, and hypertrophy will be assessed at baseline, 4 weeks, and 8 weeks. Data will be analyzed using SPSS, with appropriate parametric or non-parametric tests applied after checking data normality. Ethical approval will be obtained, informed consent will be secured, and participant confidentiality will be strictly maintained.

DETAILED DESCRIPTION:
This study is a single-blinded randomized controlled trial designed to evaluate and compare the therapeutic effectiveness of eccentric training with blood flow restriction (ECC+BFR) and heavy slow resistance (HSR) training in individuals diagnosed with chronic unilateral lateral epicondylitis. The study will be conducted at Sakina Memorial Hospital Sheikhupura and University of Lahore Teaching Hospital over a duration of 9 months following synopsis approval.

A total sample size of 40 participants (20 per group) has been determined using Epitool software, based on the Patient-Specific Functional Scale (PSFS), with a confidence level of 95%, power of 80%, and a 10% attrition allowance. Participants aged 25-45 years, of both genders, with clinically confirmed chronic lateral epicondylitis (positive Cozen's and Mill's tests) and symptom duration exceeding 12 months, will be included. Individuals with prior surgery, recent injections, systemic inflammatory conditions, vascular or clotting disorders, contraindications to BFR, pregnancy, or psychological illness will be excluded.

Eligible participants will be enrolled after providing written informed consent and randomized using a computer-generated block randomization method, with allocation concealment ensured through sealed opaque envelopes. Outcome assessors will be blinded to group allocation to minimize assessment bias.

The interventional group will receive eccentric wrist extensor exercises combined with blood flow restriction therapy, using a pneumatic cuff inflated to 50-60% limb occlusion pressure. Exercises will be performed at 20-30% 1-RM using a 30-15-15-15 repetition protocol, emphasizing slow controlled eccentric contractions. Sessions will be conducted three times weekly for 8 weeks, totaling 24 supervised sessions.

The control group will undergo a heavy slow resistance training protocol, involving wrist extensor exercises performed at 70-85% of 1-RM, with slow concentric and eccentric phases (3 seconds each). Participants will complete 3-4 sets of 6-8 repetitions, with adequate rest intervals, following the same session frequency and duration as the intervention group.

Primary and secondary outcome measures include pain intensity (Numeric Pain Rating Scale), patient-specific functional performance (PSFS), muscle strength, and muscle hypertrophy, assessed at baseline, 4 weeks, and 8 weeks post-intervention. Data will be analyzed using SPSS (version 25/27). Descriptive statistics will summarize participant characteristics, while inferential statistics will be applied based on data distribution, with significance determined accordingly.

Ethical considerations will strictly adhere to the guidelines of the Institutional Research Ethics Board (IREB), University of Lahore. Participant confidentiality, voluntary participation, right to withdraw, and safety monitoring will be ensured throughout the study. No serious adverse effects are anticipated.

ELIGIBILITY:
Inclusion Criteria:

Patient aged between 25 and 45 years. Both male and female participants with unilateral symptoms only. Clinically diagnosed unilateral lateral epicondylitis (LE), confirmed by positive Cozen's and Mills' tests. Symptom duration exceeding 12 months, indicating chronic LE.

Exclusion Criteria:

Previous history of surgery or injection therapy for LE within the past 6 months.

Coexisting conditions (e.g., rheumatoid arthritis, cervical radiculopathy, significant tendon tears). Contraindications to BFR (e.g., DVT, vascular disease, uncontrolled hypertension, clotting disorders).

Use of anticoagulants or long-term pain medications. Pregnant or psychological person.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity (Numeric Pain Rating Scale) | Baseline, 4 weeks, and 8 weeks
  Pain intensity will be assessed using the Numeric Pain Rating Scale (NPRS), a validated 11-point scale ranging from 0 (no pain) to 10 (worst imaginable pain). Participants will rate their average elbow pain during daily activities involving the affected upper limb.

SECONDARY OUTCOMES:
Patient-Specific Functional Performance (PSFS) | Baseline, 4 weeks, and 8 weeks
  Functional performance will be assessed using the Patient-Specific Functional Scale (PSFS). Participants will identify activities affected by lateral epicondylitis and rate their ability to perform each activity on an 11-point scale ranging from 0 (unable to perform) to 10 (able to perform at pre-injury level). Higher scores indicate improved functional ability.

CONTACTS AND LOCATIONS:
Overall Officials: Nimra Rafiq, MS MSK, Principal Investigator — The University of Lahore, Lahore
Locations (1):
- University of Lahore Teaching Hospital, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No